CLINICAL TRIAL: NCT06139159
Title: CRISOL Mente: A Multilevel Community Intervention to Reduce Mental Health Disparities Among Latinos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Esperanza Health Center (Unknown); The Philadelphia AIDS Consortium (Unknown)
Responsible Party: Principal Investigator, Ana Martinez Donate, Professor of Community Health and Prevention, Drexel University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MD018206 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Depression, Unipolar; Anxiety Disorders; Post Traumatic Stress Disorder
Keywords: Mental health; Latino health; Immigrant health; Community-health worker
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Intervention Model Description: Our team vision is to develop a multi-level community-based model that is more pragmatic, efficient and effective than programs that address only one level of the socioecological model or rely solely on highly trained mental health professionals, who do not always have the necessary cultural or linguistical competency and are not affordable to many Latino-serving organizations. By tackling multiple levels and domains of influence, and leveraging heavily on cultural and context concordant actors, this project can pave the way for a new, scalable, and sustainable model to improve mental health and mental health treatment among Latino communities in the U.S. The comparison of the three phases can help to identify the optimal level of involvement by the LHWs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LHW as outreach agents/navigators (Experimental): Conduct outreach activities with people in the community who are hard to reach and with limited access to health care, conduct screening for symptoms of mental illnesses, encourage and refer individuals at-risk, suspected of having, or affected by mental health issues for further triage.
  Interventions: Other: Outreach/navigator
- LHW as navigators and auxiliary to care (Experimental): LHW continue conducting outreach and referral activities but in addition, LHW are more involved in their care. They arrange consultations, introduce the patient to the clinical team via a "warm hand-off" and assist in scheduling a follow-up visit, help patients comply with the follow-up appointments, help reduce patient and system barriers impeding their care; help patients address barriers through education, referral, and navigation to ancillary community services. They have frequent contact with the patient.
  Interventions: Other: Outreach/navigator; Other: Auxiliary to care
- LHW stepped care and task shifting (Experimental): LHW conduct activities of prior arms but in addition, they may provide specific components of mental health care (task-shifting), providing components of basic evidence-based treatments to patients with non-complex needs, and addressing other syndemic health and social conditions.
  Interventions: Other: Outreach/navigator; Other: Auxiliary to care; Other: Stepped care and task shifting

INTERVENTIONS:
Other: Outreach/navigator — * Conduct outreach activities with people in the community who are hard to reach and with limited access to health care, conduct informal screening for symptoms of mental illnesses, encourage and refer individuals at-risk, suspected of having, or affected by mental health issues to clinics for triage.
  * Document outreach, screening, and referral activities in LHW database
  Other Names: Phase 1
Other: Auxiliary to care — * Arrange consultation for those at-risk, suspected, or affected individuals at clinics for triage.
  * Introduce the patient to the clinical team via a "warm hand-off" and assist in scheduling a follow -up visit.
  * Support patients in attending their clinic visits; help patients address barriers through education, referral, and navigation to ancillary community services (SAVAME, legal, housing, economic, etc);
  * Engage, activate, and empower patients to participate in the care process
  * Frequent contact with patients: +1 every two weeks during the first 3 months, +1 every month for months 4-6.
  * Assist with group sessions: affinity groups
  * Identify community-based resources.
  * Document outreach, screening, referral, and auxiliary care activities in LHW database
  Other Names: Phase 2
  Arms: LHW as navigators and auxiliary to care; LHW stepped care and task shifting
Other: Stepped care and task shifting — * Support counselling initiated by the psychologist
  * Reinforce patient education about depression, anxiety, trauma, and other syndemic conditions.
  * Work with patients' families and peers to reduce stigma, address syndemic factors and social conditions.
  * Contact frequency with patients: +1 every two weeks during the first 3 months, +1 every month for months 4-6.
  * Co-lead group sessions: affinity groups
  * Provide Mental Health First Aid to members of the community.
  * Document outreach, screening, referral, auxiliary and stepped care activities in LHW database
  Other Names: Phase 3
  Arms: LHW stepped care and task shifting

SUMMARY:
Latinos in the U.S. experience significant disparities in access to mental health services due to lack of health insurance, language barriers, low availability of bilingual providers, mental health stigma, and fear of deportation. There is an urgent need to identify low-cost, culturally appropriate interventions to reduce mental health disparities among this population. This project will address that need by implementing and testing CRISOL Mente, a multi-level, culturally-congruent community intervention to improve the mental health of the Latino population in Philadelphia.

DETAILED DESCRIPTION:
Latinos in the U.S. experience significant disparities in access to mental health services due to lack of health insurance, cost of services, limited awareness of mental health resources, mental health stigma, and fear of deportation. Limited English proficiency coupled with an acute lack of bilingual and culturally competent providers further impede Latinos' adequate access to quality mental health services. The COVID-19 pandemic has only amplified the need for mental health care and exacerbated mental health disparities for Latino communities, making it urgent to identify low-cost, effective strategies to reduce these gaps. This 5-year project seeks to develop and test a multi-level, community intervention to improve mental health outcomes and promote access to culturally appropriate mental health treatment for Latino communities in Philadelphia. CRISOL Mente will include components at various levels of the socio-ecological model: a clinic-based, stepped-care program relying on Latino lay health workers (LHW) for the delivery of mental health services.

To improve mental health symptoms and engagement in care, the investigators will recruit, train and supervise a cohort of Latino LHW who will be embedded into two Latino-serving clinics, extending the reach and effectiveness of the clinics' mental health services. The investigators will compare the impact of three different levels of LHW involvement: a) community outreach/navigation (i.e. screening and referral of community members); b) auxiliary care (i.e. screening, referral, and help overcoming barriers to better mental health); and c) task shifting (i.e. screening, referral, assistance, and supervised delivery of basic mental health treatment). The LHWs will also conduct outreach/education activities in the community (e.g. radio talks, info sessions, tables in community venues) to reduce mental health stigma. Our experienced and largely Latino community-academic research team will also engage in capacity building activities (i.e. monthly town halls, annual retreats, weekly newsletters, provision of trainings and technical support) with the Latino Health Collective, a coalition of Latino-serving organizations. Using mixed-methods and the RE-AIM framework, CRISOL Mente's impact will be evaluated with clinical data, baseline and 6-month patient survey data (N=200 from each level of LHW involvement, total n=600).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Fluent in English or Spanish
* Self-identification as a member of the Latino community
* Resident of Philadelphia, Bucks, Montgomery, Delaware, or Chester County.
* Moderate to severe clinical symptoms of anxiety, depression, and/or PTSD

Exclusion Criteria:

* People with high-risk mental health symptoms: active suicidality, substance use disorder, mania, psychosis, and schizophrenia
* People already receiving mental health therapy (in the last 3 months)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in mental health symptomatology (depressive, anxiety or post-traumatic stress disorder [PTSD]) | Baseline to 6 months
  Improvement is a composite measure defined as change in any of the mental health outcomes. The following scales and categories will be used to define improvement.
  * Depressive symptoms: decrease in from CESD-10 at bsl >=10 to CESD-10 <10 at 6-month, among those with CESD-10 >=10 at baseline, OR
  * Anxiety symptoms: decrease in GAD7 category from bsl to 6-month: from 15-21(severe) to 10-14 (moderate) or from 15-21(severe) to less than 10 (mild or minimal anxiety), or from 10-14 bsl (moderate) to less than 10 (mild or minimal anxiety), among those with GAD7 >=10 at baseline, OR
  * For PTSD, decrease from in PTSD category from bsl to 6 months: from >=3 to PTSD <3, among those with PTSD>=3 at baseline).

SECONDARY OUTCOMES:
Depressive symptomatology | Baseline to 6 months
  Presence or absence of any clinical mental health disorder will be determined using Center for Measured using Epidemiologic Studies Depression Scale Revised (CESD-R10) for depressive symptoms (continuously)
Anxiety symptomatology | Baseline to 6 months
  Measured using General Anxiety Disorder-7 (GAD-7) scale for anxiety symptoms (continuosly)
Post traumatic stress disorder symptomatology | Baseline to 6 months
  Measured using the Short Screening Scale for post-traumatic stress disorder (PTSD).

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University School of Public Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No